CLINICAL TRIAL: NCT00076687
Title: Safety Study of Botulinum Toxin Type A in Post-Upper Limb Stroke Patients With Reduced Lung Function
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 191622-057
Record Dates: First submitted 2004-01-29; First posted 2004-02-26 (Estimated); Results first posted 2011-10-03 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-08

CONDITIONS: Stroke; Muscle Spasticity; Motor Neuron Disease
MeSH Terms: conditions — Stroke; Muscle Spasticity; Motor Neuron Disease | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental)
  Interventions: Biological: botulinum toxin Type A
- 2 (Experimental)
  Interventions: Biological: botulinum toxin Type A
- 3 (Placebo Comparator)
  Interventions: Drug: saline

INTERVENTIONS:
Biological: botulinum toxin Type A — botulinum toxin Type A 240 U injection on Day 1, Week 12, Week 18
  Other Names: BOTOX®
  Arms: 1
Biological: botulinum toxin Type A — botulinum toxin Type A 360 U injection at Day 1, Week 12, Week 18
  Other Names: BOTOX®
  Arms: 2
Drug: saline — Saline injection at Day 1, Week 12, Week 18
  Arms: 3

SUMMARY:
The purpose of this study is to evaluate the safety of injections of botulinum toxin Type A in patients with reduced lung function and focal upper limb poststroke spasticity

ELIGIBILITY:
Inclusion Criteria:

* Abnormal pulmonary function test results;
* focal, upper limb spasticity, upper motor neuron syndrome

Exclusion Criteria:

* Previous exposure to botulinum toxin of any serotype

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2003-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (4):
- Miami, Florida, United States
- Prague, Czechia
- Szeged, Hungary
- Warsaw, Poland

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
- Botulinum Toxin Type A 240 U: botulinum toxin Type A 240 U
- Botulinum Toxin Type A 360 U: botulinum toxin Type A 360 U
Period: Overall Study
Arm/Group | Placebo | Botulinum Toxin Type A 240 U | Botulinum Toxin Type A 360 U
Started | 48 | 52 | 55
Completed | 42 | 47 | 51
Not Completed | 6 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Botulinum Toxin Type A 240 U | Botulinum Toxin Type A 360 U | Total
Number analyzed (Participants) | 48 | 52 | 55 | 155
Age Continuous [Mean (Full Range); unit: years] | 58 [18 to 80] | 55.5 [21 to 83] | 55.8 [19 to 81] | 56.4 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 13 | 21 | 53
  Male | 29 | 39 | 34 | 102

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Vital Capacity (FVC)
Description: Change from baseline in observed FVC. FVC is the maximum amount of air exhaled from the lungs after taking the deepest breath possible. Patients perform three to eight exhalations into a spirometer with the highest value recorded at Baseline and Week 6.
Time Frame: Baseline, Week 6
Population: Safety
Measure: Mean (Standard Deviation); unit: Liters of air
Arm/Group | Placebo | Botulinum Toxin Type A 240 U | Botulinum Toxin Type A 360 U
Number analyzed (Participants) | 48 | 52 | 55
Liters of air
  Baseline | 2.889 (0.7804) | 3.068 (0.8766) | 2.923 (0.7627)
  Change from Baseline at Week 6 | 0.057 (0.3151) | 0.052 (0.2883) | -0.081 (0.2531)

2. Primary Outcome: Change From Baseline in Forced Expiratory Volume (FEV1)
Description: Change from baseline in observed FEV1 at one second. FEV1 is the maximum amount of air exhaled in one second. Patients perform three to eight exhalations into a spirometer with the highest value recorded at Baseline and Week 6.
Time Frame: Baseline, Week 6
Population: Safety
Measure: Mean (Standard Deviation); unit: Liters of air
Arm/Group | Placebo | Botulinum Toxin Type A 240 U | Botulinum Toxin Type A 360 U
Number analyzed (Participants) | 48 | 52 | 55
Liters of air
  Baseline | 2.111 (0.5944) | 2.223 (0.6492) | 2.168 (0.6568)
  Change from Baseline at Week 6 | 0.049 (0.1971) | 0.023 (0.2925) | -0.008 (0.2340)

3. Secondary Outcome: Change From Baseline in FEV1/FVC Ratio
Description: Change from baseline in FEV1/FVC ratio. This ratio is calculated by dividing the FEV1 value by the FVC value. This represents that portion (or ratio) of FVC exhaled in one second.
Time Frame: Baseline, Week 6
Population: Safety
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo | Botulinum Toxin Type A 240 U | Botulinum Toxin Type A 360 U
Number analyzed (Participants) | 48 | 52 | 55
Ratio
  Baseline | 0.741 (0.1320) | 0.731 (0.1260) | 0.742 (0.1051)
  Change from Baseline at Week 6 | 0.000 (0.0730) | -0.006 (0.0709) | 0.019 (0.0699)

4. Secondary Outcome: Change From Baseline in Ashworth Scale
Description: Change from Baseline in worst upper limb scores using the Ashworth Scale at Week 6 from Baseline. Upper limb includes finger, wrist, thumb, and elbow. Worst score was the highest value measured from the finger, wrist, thumb, or elbow at Baseline and Week 6 based on treated areas. The Ashworth Scale assesses the degree of muscle tone. It is a 5-point scale where 0 equals no increase in muscle tone and 4 equals very severe muscle rigidity. A low score indicates little or no stiffness. A high score indicates severe stiffness. A negative change from baseline score indicates improvement.
Time Frame: Baseline, Week 6
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: Number on a scale
Arm/Group | Placebo | Botulinum Toxin Type A 240 U | Botulinum Toxin Type A 360 U
Number analyzed (Participants) | 48 | 52 | 55
Number on a scale
  Baseline | 3.19 (0.607) | 2.87 (0.561) | 2.96 (0.693)
  Change from Baseline at Week 6 | -0.60 (0.564) | -1.01 (0.801) | -1.16 (0.834)

ADVERSE EVENTS:
Arm/Group | Placebo | Botulinum Toxin Type A 240 U | Botulinum Toxin Type A 360 U
Serious Adverse Events (participants affected / at risk) | 7/48 | 9/52 | 6/55
Other Adverse Events (participants affected / at risk) | 18/48 | 15/52 | 17/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | Botulinum Toxin Type A 240 U (N=52) | Botulinum Toxin Type A 360 U (N=55)
Abscess (Infections and infestations) | 0 | 1 | 0
Acute endocarditis (Infections and infestations) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Splenic abscess (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 2
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Encephalitis (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Meningocele (Congenital, familial and genetic disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 1
Heart rate decreased (Investigations) | 0 | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=48) | Botulinum Toxin Type A 240 U (N=52) | Botulinum Toxin Type A 360 U (N=55)
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 2
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3 | 2
Headache (Nervous system disorders) | 3 | 0 | 3
Muscle spasticity (Nervous system disorders) | 0 | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.